CLINICAL TRIAL: NCT00818480
Title: Phase II: An Open-Label Extension Study of 168-Hour Continuous Infusion of YM155 in Subjects Previously Enrolled in a Phase I or Phase II Protocol Administering YM155
Brief Title: An Extension Study Administering YM155 to Subjects Previously Enrolled in Another Protocol Administering YM155
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-101
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Prostate Cancer; Melanoma; Non-Hodgkin's Lymphoma
Keywords: prostate cancer; melanoma; lymphoma; YM155
MeSH Terms: conditions — Prostatic Neoplasms; Melanoma; Lymphoma, Non-Hodgkin; Lymphoma | interventions — sepantronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1. YM155 (Experimental)
  Interventions: Drug: YM155

INTERVENTIONS:
Drug: YM155 — continuous infusion

SUMMARY:
This protocol is open to subjects previously enrolled in and who had completed a Phase I or Phase II study administering YM155. Subjects who are receiving benefit from treatment with YM155 are eligible after completing the previous study.

DETAILED DESCRIPTION:
The main objective of the study is to continue to evaluate the safety and efficacy of YM155.

Each subject will be treated at the dose he/she was receiving at the completion of his/her previous phase I or phase II YM155 study.

ELIGIBILITY:
Inclusion Criteria:

* Completed a Phase I or II YM155 study with at least stable disease and continues to meet the criteria as stated in the previous YM155 study that allows for additional treatment with YM155
* Lack of progression based on the most recent radiological imaging, biochemical assessments and/or physical examination
* Negative pregnancy test result (females of child-bearing potential)

Exclusion Criteria:

* More than 21 days (or 14 days depending on the study of origin) between the time the last infusion of YM155 was stopped in the previous study and the proposed start of the first infusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02; Primary Completion 2011-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Assess Response Rate | End of Study up to 77 months
Safety assessed by recording of adverse events, physical examinations, vital signs, laboratory assessments and electrocardiograms (ECGs) | End of Study up to 77 months

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director, Study Director — Astellas Pharma Global Development
Locations (3):
- United States (3):
  - Institute for Drug Development, San Antonio, Texas
  - South Texas Accelerated, San Antonio, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah